CLINICAL TRIAL: NCT02419352
Title: Effect of Sugammadex Versus Neostigmine/Atropine Combination on Cognitive Function After Elective Adult Surgery
Brief Title: Sugammadex and Cognitive Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, Chrysanthi Batistaki, Assistant Professor of Anesthesiology, 2nd Department of Anesthesiology, School of Medicine, University of Athens, Attikon Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 331/21-9-10
Record Dates: First submitted 2015-04-08; First posted 2015-04-17 (Estimated); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Post Operative Cognitive Dysfunction
Keywords: Cognitive function
MeSH Terms: interventions — Sugammadex; Neostigmine; Atropine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sugammadex (Active Comparator): Sugammadex is administered to reverse rocuronium-induced neuromuscular blockade at the end of elective surgery.
  Interventions: Drug: Sugammadex
- Neostigmine/atropine (Active Comparator): Neostigmine combined to atropine is administered to reverse rocuronium-induced neuromuscular blockade at the end of elective surgery.
  Interventions: Drug: Neostigmine/atropine

INTERVENTIONS:
Drug: Sugammadex
  Other Names: Bridion
  Arms: Sugammadex
Drug: Neostigmine/atropine
  Arms: Neostigmine/atropine

SUMMARY:
Post operative cognitive dysfunction (POCD) is recognized as a frequent complication after both cardiac and non cardiac surgery, affecting approximately 1/3 of the patients. The aim of this study is to examine the possible effect of the novel reversal agent sugammadex versus neostigmine/ atropine combination on cognitive function of adult patients after elective surgery during the early post operative period as well as at discharge.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >40 years old
* ASA I-III
* Patients scheduled for elective surgery with general anaesthesia.

Exclusion Criteria:

* Neuro-, vascular-, orthopedic- or cardiac surgery
* Known psychiatric or disease of the CNS
* History of craniotomy
* Receiving tranquillisers or antidepressants on a regular basis pre-operatively
* Alcoholism or drug dependence
* History of stroke
* Refusal of patient
* Inability to read or write
* MMSE < 22 pre-operatively

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2010-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in the Mini-Mental State Evaluation test | Preoperatively, 1 hour postoperatively, at discharge (1-15 days postoperatively)
Change in the clock-drawing test | Preoperatively, 1 hour postoperatively, at discharge (1-15 days postoperatively)
Change in the Isaacs set test | Preoperatively, 1 hour postoperatively, at discharge (1-15 days postoperatively)

SECONDARY OUTCOMES:
Time from reversal agent administration to extubation | After reversal agent administration

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Department of Anesthesiology, Attikon Hospital, 1 Rimini str., Athens, Greece